Universitat Internacional de Catalunya



## **INFORMED CONSENT FORM**

Study Number: FIS-2020-02

Protocol version: 1.0 Date: 08.07.2020

Research title: Using the App as a guide to lumbopelvic stability exercises in patients with chronic stroke: a

pilot study of a randomized clinical trial

Universitat Internacional de Catalunya

Comitè d'Ètica d'Investigació amb medicaments



| I, Mr./Mrs .: | |
|---|---|
| <ul> <li>I have received verbal information about the study and have r<br/>which I have received a copy.</li> </ul> | read the attached written information, of |
| <ul> <li>I have understood what has been explained to me.</li> </ul> | |
| <ul> <li>I have been able to make comments about the study and ask</li> <li>I give my consent to take part in the study and I assume that n</li> <li>I understand that I may withdraw at any time without affecting</li> </ul> | my participation is completely voluntary. |
| By signing this informed consent form, I give my consent so that my print in this consent form, which complies with the provisions of Organic Law Personal Data and guarantee of digital rights | |
| I understand that I will receive a copy of this informed consent form. | |
| Signature of the patient or the patient | Signature Date |
| ID number | |
| STATEMENT OF THE INVESTIGATOR OR INVESTIGATOR | |
| The patient or patient who signs this consent form has received, from oral and written form of the process and nature of this research study, questions regarding the nature, the risks and benefits of participating in | and has had the opportunity to ask any |
| Signature of the researcher Name: | Fecha de la firma |